CLINICAL TRIAL: NCT02401607
Title: SEEK Study - Study on Emergency Health Care Workers' Job Strain Evaluated by Karasek Questionnaire
Acronym: SEEK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Association des Médecins des Urgences de Clermont-Ferrand (Other); Université d'Auvergne (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0228
Record Dates: First submitted 2015-03-16; First posted 2015-03-30 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Health Care Workers
Keywords: emergency Medecine; biomarkers of stress; Food intake

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Karasek questionnaire and Saliva prelevement — Karasek questionniare and Saliva collection will be assessed on any health care worker working in any emergency department in France at day 1 and at 5 years

SUMMARY:
Emergency health care workers are exposed to job strain - defined by Karasek as a combination of high job demands and low job control. Emergency health care work is a complex interaction between stress due to life-threatening emergencies, overcrowding of the Emergency Department, the lack of sleep, bad food repartition during shifts, and accumulated fatigue. However, the Karasek questionnaire has never been assessed for Emergency Health Care workers. Furthermore, the variation of results during the career has never been assessed.

The same measures will be repeated every 5 year to assess long term changes in subjective and objective measures of stress.

The study's main objective is the creation of an Emergency Health Care worker's cohort to assess the evolution of the Karasek questionnaire during the follow-up.

Secondary objectives are

* the evaluation of the food intake before, during and after a nightshift.
* the evaluation of other questionnaires

DETAILED DESCRIPTION:
Chronic stress at work is a public health problem increasing morbidity and mortality. Emergency physicians is particularly an at risk population. Indeed, their work is a complex interaction between stress due to life-threatening emergencies, the lack of sleep and accumulated fatigue.

A way of measuring stress at work is the use of self-reported psychological questionnaire. Among them, the Job control demand model from Karasek is widely used to evaluate psychosocial factors at work. The Karasek job strain model has been assessed in 25 000 workers in the Sumer study and allowed to classify the main types of occupations. However, no data regarding emergency physicians scores at the Karasek questionnaire were available, even though burnout exposure is a well-known problematic among health care workers. This absence is particularly unfortunate as emergency physicians often needs to deals with life threatening emergency in a short amount of time, following regularly long and craving shifts. A preliminary study with a low sample size reported in concrete terms the atypical "out of limit" situations of emergency physicians, with a decision latitude among the lowest and the highest psychological demand ever reported. Moreover, variation of stress at work has been linked with professional experiences. Karasek questionnaire is supposed to assess a long-term stable perception of work, despite the absence of study comparing Karasek scores within different conditions in the same participant. It is also important to explore protective factors that might help alleviate perceived stress and that are quite easy to integrate into medical organizations or in daily lifestyle.

Finally, several biomarkers of stress have been proposed. Among them, our team previously highlighted the potential of DHEAS to assess stress, due to its stability (steroid) and its long half-life of 16 hours. To our knowledge, the relationships between biomarkers of stress and the Karasek job strain model have never been investigated. Comparisons between emergency health care workers are also lacking.

Therefore, the general aim of this study is to enhance psychological well-being in emergency physicians. The primary objective is to verify our preliminary findings at Karasek scores on a large sample size of emergency physicians. The secondary objectives are to evaluate whether there is a change in perception of work both at short-term (on leave and after a 24-hour shift) and long-term (with professional experience). We will further explore its relationships with some biomarkers of stress and protective factors. Moreover, we aim to compare emergency health care workers specificity.

Questionnaires and saliva collection will be performed twice: at the beginning of a day work and at the end of a night work. Both measures will be recorded at the same time within each participant, between 6.30 am and 8.30 am depending of the health care workers. The time required by participant is evaluated to about 15min each time.

The same measures will be repeated every 5 year to assess long term changes in subjective and objective measures of stress.

The population description will be achieved with descriptive statistics. Continuous variables will be presented as mean and standard deviation, under the normality of distribution condition (Shapiro-Wilk needed).

The primary analysis will be mainly descriptive and will express (as a quantitative and categorical variables) the perception scores of emergency physicians work according to the Karasek questionnaire, for each dimensions composing the score (decision latitude, psychological demands and social support).

The evolution of the Karasek questionnaire score, obtained for each dimension, will be tested with a paired two-sample emergency physician's test (or nonparametric Wilcoxon test if necessary). Linear regression models or aleatory effects models (as described by Klar and Darlington, 2004, in Statistics in Medicine) will eventualy complete these analyzes. This will permit, with multivariate analyzes and the introduction of covariates, to seek for possible explanatory factors of the Karasek score and its evolution. The same process will be used for quantitative parameters that will be collected.

All statistical analyses will be performed as bilateral tests with a p <0.05 considered as significant. Statistical analyzes will be performed using STATA 16 software (Stata Corporation, College Station).

ELIGIBILITY:
Inclusion Criteria:

* Any health care workers from any emergency department of France

Exclusion Criteria:

* Pregnancy
* Refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: health care workers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Karasek questionnaire | at day 1
  Karasek questionnaire is a self-reported psychological questionnaire. It defines job demands and job control as the two broad work-related characteristics present in the environment of most occupations that can be incredibly stressful. Workers can perceive both job demand and job control as being low or high. The combination of high job demands and low job control results in "Job Strain"
Karasek questionnaire | at 5 years
  Karasek questionnaire is a self-reported psychological questionnaire. It defines job demands and job control as the two broad work-related characteristics present in the environment of most occupations that can be incredibly stressful. Workers can perceive both job demand and job control as being low or high. The combination of high job demands and low job control results in "Job Strain"
Karasek questionnaire | at 10 years
  Karasek questionnaire is a self-reported psychological questionnaire. It defines job demands and job control as the two broad work-related characteristics present in the environment of most occupations that can be incredibly stressful. Workers can perceive both job demand and job control as being low or high. The combination of high job demands and low job control results in "Job Strain"

SECONDARY OUTCOMES:
Hamilton anxiety scale | at day 1, at 5 years, 10 years
  It is a psychological questionnaire used by clinicians to rate the severity of a patient anxiety.
Maslach Burn-out Inventory | at day 1, at 5 years, 10 years
  It is a psychological assessment instrument comprising 22 symptom items pertaining to occupational burnout.
Hospital anxiety and depression scale | at day 1, at 5 years, 10 years
  It is used by doctors to determine the levels of anxiety and depression that a person is experiencing
Assessment of the food intake | at day 1
  Questionnaire created by our team to assess the quantitative and qualitative food intake before, during and after a nightshift.
Assessment of the salivary DHEA levels | at day 1
  Salivary DHEA is a biomarker of stress

CONTACTS AND LOCATIONS:
Overall Officials: Frederic DUTHEIL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Bouillon-Minois JB, Trousselard M, Pereira B, Schmidt J, Clinchamps M, Thivel D, Ugbolue UC, Moustafa F, Occelli C, Vallet G, Dutheil F. Protocol of the Study on Emergency Health Care Workers' Responses Evaluated by Karasek Questionnaire: The SEEK-Study Protocol. Int J Environ Res Public Health. 2021 Apr 12;18(8):4068. doi: 10.3390/ijerph18084068. PMID 33921527